CLINICAL TRIAL: NCT02304601
Title: Entwicklung Und Testung Eines Generischen Screenings für Die Vorabschätzung Von Fallgruppen im Antragsverfahren
Brief Title: Development and Testing of a Generic Screening for Use in Application Process of Medical Rehabilitation Services
Acronym: Generik
Status: Completed | Type: Observational
Sponsor: Martin Brünger (Other)
Collaborators: Deutsche Rentenversicherung (Other)
Responsible Party: Sponsor-Investigator, Martin Brünger, M.D., MPH, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: 8011-106-31/31.27.16
Record Dates: First submitted 2014-11-25; First posted 2014-12-02 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2014-11

CONDITIONS: Medical Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Comorbid symptoms
- No comorbid symptoms

SUMMARY:
The primary objective of this research is the development and testing of a brief cross-indication instrument (screening) for use in the approval process of medical rehabilitation services. In addition to the empirical foundation, this generic instrument should have a high level of acceptance of both applicants and payers of rehabilitation services. Furthermore, an everyday and economic use for the routine application process for medical rehabilitation services at the German statutory pension insurance scheme should be provided. In the first study phase, a long instrument was tested with a sample of rehabilitees that received approval of medical rehabilitation services. This assessment including the measurement of rehabilitation-related somatic, psychological and social impairments was first tested for its psychometric properties and then reduced to a short instrument (screening) using quantitative methods. In the second study phase, the then-existing screening will be part of the application documents for medical rehabilitation services to assess its management properties and practicability in everyday use of the German statutory pension insurance scheme.

ELIGIBILITY:
Inclusion Criteria:

* Member of German Federal Pension Insurance
* Approval of a medical rehabilitation according to § 15 SGB VI

Exclusion Criteria:

* Returning questionnaire after beginning of medical rehabilitation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the German Federal Pension Insurance before their medical rehabilitation
Sampling Method: Probability Sample
Enrollment: 2736 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
return-to-work | up to 9 months
  The outcome is assessed by the discharge report from the rehabilitation centre.

SECONDARY OUTCOMES:
therapies during rehabilitation | up to 9 months
  The outcome is assessed by the discharge report from the rehabilitation centre according to the 'classification of therapeutical services'.
socio-medical prognosis | up to 9 months
  The outcome is assessed by the discharge report from the rehabilitation centre.

REFERENCES:
- [Background] Streibelt M, Brunger M. [How many work-related therapeutic services do patients with severe restrictions of work ability receive? Analysis of a representative rehabilitation sample across indications]. Rehabilitation (Stuttg). 2014 Dec;53(6):369-75. doi: 10.1055/s-0034-1375643. German. PMID 25185025
- [Background] Brunger M, Spyra K. Prevalence of comorbid depressive symptoms in rehabilitation: A cross-indication, nationwide observational study. J Rehabil Med. 2016 Nov 11;48(10):903-908. doi: 10.2340/16501977-2156. PMID 27735981
- [Result] Brunger M, Streibelt M, Schmidt C, Spyra K. [Psychometric Testing of a Generic Assessment Tool for the Identification of Biopsychosocial Impairments in Persons with an Approval for Medical Rehabilitation]. Rehabilitation (Stuttg). 2016 Jun;55(3):175-81. doi: 10.1055/s-0042-104668. Epub 2016 Jun 10. German. PMID 27284731